CLINICAL TRIAL: NCT06070831
Title: Comparison Between Two Respiratory Muscle Training Protocols: Inspiratory Muscle Training vs Expiratory Muscle Training in Acquired Brain Injury Patients.
Brief Title: Respiratory Muscle Training in Acquired Brain Injury Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, CARLOS MARTIN SANCHEZ, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23092023
Record Dates: First submitted 2023-09-23; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Disease; Muscle Weakness; Acquired Brain Injury; Older People--Abuse of; Physical Inactivity
MeSH Terms: conditions — Respiration Disorders; Muscle Weakness; Brain Injuries; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The professional that collected the data and the participants were unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (IMT) (Experimental): Inspiratory muscle training at 50% of MIP, the training load was set each 2 weeks to keep 50% of MIP.
  Interventions: Device: Inspiratory muscle training
- Expiratory muscle training group (EMT) (Experimental): Expiratory muscle training at 50% of MEP, following the same rules as HIT.
  Interventions: Device: Expiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Respiratory training, performed through IMT, was carried out with a pressure threshold device (Treshold IMT, Philips-Respironics, Pittsburg, PA, USA). Threshold IMT offers a constant and specific pressure for strength and endurance training of the respiratory muscles, regardless of the strength or speed with which patient breathes. A flow-independent one-way valve ensures constant resistance and allows you to specifically adjust workload (in cmH2O). The training must be supervised by a healthcare professional. During the inspiration, a spring-loaded valve resists to stimulate the training of the respiratory muscles. Before training began, the participants and primary caregivers completed one-session familiarization with a specialist to know the operation of the device.
  Adult people with acquired brain injury carried out the training program for 8 weeks, 1 session every day, 5 days a week. The participants performed 5 series of 1 minute with 1-minute rest between them.
  Arms: Inspiratory muscle training group (IMT)
Device: Expiratory muscle training — Respiratory training, performed through PEP, was carried out with a pressure threshold device (Treshold PEP, Philips-Respironics, Pittsburg, PA, USA). Threshold PEP offers a constant and specific pressure for strength and endurance training of the respiratory muscles, regardless of the strength or speed with which patient breathes. A flow-independent one-way valve ensures constant resistance and allows you to specifically adjust workload (in cmH2O). The training must be supervised by a healthcare professional. During the expiration, a spring-loaded valve resists to stimulate the training of the respiratory muscles. Before training began, the participants and primary caregivers completed one-session familiarization with a specialist to know the operation of the device.
  Adult people with acquired brain injury carried out the training program for 8 weeks, 1 session every day, 5 days a week. The participants performed 5 series of 1 minute with 1-minute rest between them.
  Arms: Expiratory muscle training group (EMT)

SUMMARY:
Background: Respiratory health problems are one of the main causes of morbidity and mortality in adult people with acquired brain injury (ABI). The influence of respiratory muscle training has not yet been studied in this population group. The objective of the study was to evaluate and compare the efficacy of two protocols with respiratory muscle training, inspiratory muscle training vs expiratory muscle training, to improve respiratory strength and pulmonary function in adults with CP.

Methods: The study is a controlled, randomised, double-blind trial and with allocation concealment. 26 ABI patients will be recruited and randomly distributed in the inspiratory muscle training group (IMT) and the expiratory muscle training group (EMT). Over an 8-week period an IMT or EMT protocol was followed 5 days/week, 5 series of 1-minute with 1-minute rest between them. IMT trained with a load of 50% of the maximum inspiratory pressure (MIP) and EMT with 50% of the maximum expiratory pressure (MEP). Respiratory strength and pulmonary function were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Belong to ASDACE.
* Sign the Informed consent.

Exclusion Criteria:

The presence of a respiratory disease in the previous month, inability to understand assessment tests or intervention or hemodynamic alterations (heart rate > 150 beats per minute (bpm), systolic blood pressure > 140 millimeters mercury (mmHg) or diastolic blood pressure > 90 mmHg).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-12-21 (Estimated); Primary Completion 2024-02-21 (Estimated); Study Completion 2024-04-21 (Estimated)

PRIMARY OUTCOMES:
Inspiratory muscle strength | 8 weeks.
  It was measured using the maximum inspiratory pressure (MIP) with a pressure measurer (Elka PM-15, Laboliser, S.A., Barcelona, Spain), from residual volume and total lung capacity. Unit of measure, centimeter of water (cmH2O).
Expiratory muscle strength | 8 weeks.
  It was measured using the maximum expiratory pressure (MEP) with a pressure measurer (Elka PM-15, Laboliser, S.A., Barcelona, Spain), from residual volume and total lung capacity. Unit of measure, centimeter of water (cmH2O).

SECONDARY OUTCOMES:
Pulmonary volume. | 8 weeks.
  Forced expiratory volume in 1 second (FEV1). It was measured using the peak flow device (Asma-1, Vitalograph Ltd, Buckingham, England). Unit of measure, liters (L).
Pulmonary flow. | 8 weeks.
  Peak expiratory flow (PEF). It was measured using the peak flow device (Asma-1, Vitalograph Ltd, Buckingham, England). Unit of measure, liters per minute (L/min).

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS MARTIN SANCHEZ, PHD, Principal Investigator — University of Salamanca

IPD SHARING:
Plan to Share IPD: No